CLINICAL TRIAL: NCT05228613
Title: A Phase I, Observer-Blind, Randomized, Controlled Study of the Safety and Immunogenicity of SARS-CoV-2 Protein Subunit Recombinant Vaccine (Adjuvanted With Alum+CpG 1018) in Healthy Populations Aged 18 Years and Above in Indonesia
Brief Title: Safety and Immunogenicity Study of COVID-19 Protein Subunit Recombinant Vaccine Adjuvanted With Alum+CpG 1018
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other); Faculty of Medicine, Diponegoro University, Semarang (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CoV2-0122
Record Dates: First submitted 2022-02-07; First posted 2022-02-08 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; healthy population
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Observer blind: Investigational Product and Active Comparator are masking. Lot number is masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Vaccine Candidate Formula A (Experimental): 2 doses of vaccine candidate formula A administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 protein subunit recombinant vaccine
- Vaccine Candidate Formula B (Experimental): 2 doses of vaccine candidate formula B administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 protein subunit recombinant vaccine
- Vaccine Candidate Formula C (Experimental): 2 doses of vaccine candidate formula C administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 protein subunit recombinant vaccine
- Vaccine Candidate Formula D (Experimental): 2 doses of vaccine candidate formula D administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 protein subunit recombinant vaccine
- Active Control (Active Comparator): 2 doses of active control administered with 28 days interval (0.5 mL per dose)
  Interventions: Biological: SARS-CoV-2 inactivated vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 protein subunit recombinant vaccine — candidate vaccine manufactured by PT. Bio Farma
  Arms: Vaccine Candidate Formula A; Vaccine Candidate Formula B; Vaccine Candidate Formula C; Vaccine Candidate Formula D
Biological: SARS-CoV-2 inactivated vaccine — active control manufactured by Sinovac Life Sciences Co.Ltd
  Arms: Active Control

SUMMARY:
The study is an observer-blind, randomized, controlled prospective intervention study of Phase I. The primary objective is to evaluate the safety and immunogenicity of the SARS-CoV-2 protein subunit recombinant vaccine adjuvanted with Alum+CpG1018

DETAILED DESCRIPTION:
This trial is observer blinded, comparative, randomized, phase I study. Approximately 175 subjects will be recruited (18 years and above).

The investigational product is 0.5 ml in two dose-regimen (for all subjects) with 28 days apart between doses, compare to an active control (inactivated SARS-CoV-2 vaccine). There will be 4 formula of investigational product used with different concentration of Receptor Binding Domain (RBD) antigen and adjuvant CpG 1018.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy subjects aged 18 years and above.
2. Subjects have been informed properly regarding the study and signed the informed consent form.
3. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. History of vaccination with any investigational product against COVID-19 (based on anamnesis)
3. Subjects who have history of COVID-19 (based on anamnesis or other examinations).
4. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. The result of RT-PCR test for SARS-CoV-2 is positive.
6. Women who are lactating, pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
7. Abnormality hematology and biochemical test results (for main study subset).
8. History of asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
9. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
10. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
11. Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
12. Subjects who have history of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome.
13. Subjects receive any vaccination (other than COVID-19 vaccine) within 1 month before and after IP immunization.
14. Subjects plan to move from the study area before the end of study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Safety of the vaccine within 7 days after each dose | 7 days after each dose
  percentage of subjects with solicited and unsolicited Adverse Events (AE)

SECONDARY OUTCOMES:
safety of the vaccine within 28 days after each dose | 28 days after each dose
  percentage of subjects with solicited and unsolicited AE
Serious Adverse Event (SAE) of the vaccine | 6 months after the last dose
  percentage of subjects with at least 1 SAE
Comparison of safety between vaccine and active control | 28 days after each dose and 6 months after the last dose
  percentage of subjects with AE and SAE between vaccine and active control group
Deviation of laboratory evaluation | 7 days after the first dose and 14 days after the last dose
  Any deviation from routine laboratory evaluation that probably related to the dosing
Inflammatory factor evaluation | 7 days after the first dose and 14 days after the last dose
  The change of interleukin-6 (IL-6) in serum
Immunogenicity profile after the last dose | 14 days and 28 days after the last dose
  GMT of IgG antibody and neutralization antibody
Immunogenicity profile after the last dose | 14 days and 28 days after the last dose
  seroconversion rate of IgG antibody and neutralization antibody
Comparison of immunogenicity profile | 14 days and 28 days after the last dose
  GMT of IgG antibody and neutralization antibody
Comparison of immunogenicity profile | 14 days and 28 days after the last dose
  seroconversion rate of IgG antibody and neutralization antibody

OTHER OUTCOMES:
Cellular immunity evaluation | 14 days after the last dose
  Positive rate of specific T-cell response

CONTACTS AND LOCATIONS:
Overall Officials: Prof Rini Sekartini, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Yetty Movieta Nency, MD, Principal Investigator — Faculty of Medicine, Diponegoro University, Semarang
Locations (2):
- Indonesia (2):
  - Faculty of Medicine, Diponegoro University, Semarang, Semarang, Central Java
  - Fakultas Kedokteran Universitas Indonesia, Jakarta, Greater Jakarta